CLINICAL TRIAL: NCT04097340
Title: Attention Training on Smartphones (The ATS Study)
Brief Title: Attention Training on Smartphones
Acronym: ATS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left Institution
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IRB201800947; OCR19813 (Other: UF OnCore)
Record Dates: First submitted 2019-09-05; First posted 2019-09-20 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Attention; Substance Use
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Attentional Training Group (Active Comparator): Each condition involves use of a smartphone app. One smartphone app includes a task that targets attention directed to substance-related cues while the other app includes a similar task that does not target attention in this way. Neither participant nor the staff members working on the study will know which condition the participant has been randomly assigned to.
  Interventions: Device: Attentional Bias Retraining (ABR)
- Control Training Group (Placebo Comparator): Each condition involves use of a smartphone app. One smartphone app includes a task that targets attention directed to substance-related cues while the other app includes a similar task that does not target attention in this way. Neither participant nor the staff members working on the study will know which condition the participant has been randomly assigned to.
  Interventions: Device: Control Training

INTERVENTIONS:
Device: Attentional Bias Retraining (ABR) — Participants randomized to this intervention will receive 2 weeks of ABR for opioids delivered via a mobile device.
  Arms: Attentional Training Group
Device: Control Training — Participants randomized to this intervention will receive 2 weeks of training without ABR, delivered via a mobile device.
  Arms: Control Training Group

SUMMARY:
The goal of this study is to evaluate a new method that may influence attention, cravings and substance use called attention training, which will be delivered on a smartphone through an application (app). The study team would like to know what participants think of this new method and to determine if research involving this app is feasible. Eligible participants will use the app for a period of two weeks and attend a total of 4 appointments at our study location.

DETAILED DESCRIPTION:
The goal of this study is to evaluate a new method that may influence attention, cravings and substance use called attention training, which will be delivered on a smartphone through an application (app). The study team would like to know what participants think of this new method and to determine if research involving this app is feasible. Eligible participants will use the app for a period of two weeks and attend a total of 4 appointments at our study location. A primary aim of the study is to assess feasibility, usability and acceptability of mobile Attention Bias Retraining (ABR) by quantifying adherence (in lab and natural environment), self-reported ease of use, perceived value and likelihood of future use. Another primary aim of the study is to determine if ABR reduces attentional bias (AB) for opioids in those with Opioid Use Disorders (OUD) compared to a control training condition. A secondary aim of the study is to assess whether ABR reduces opioid craving to a greater extent than a control training condition based on self-report. Another secondary aim is to assess whether ABR is associated with less opioid use during the training period than a control training condition based on self-report and urinalysis. An exploratory aim of the study is to measure levels of self-reported pain pre- and post- ABR. Another exploratory aim is to examine the durability of ABR effect on AB/craving/ opioid use at 1-month follow-up.

Interested individuals will first complete a in-person screening appointment including a medical and psychiatric screening and questionnaires covering topics including substance and alcohol use, cigarette smoking, and sexual behaviors. Eligible participants who enroll in the study will next complete an orientation appointment when study staff will teach participants how to use the study app and answer any questions that arise. Participants will then be randomly assigned (like a flip of a coin) to one of two conditions. Each condition involves use of a smartphone app. One smartphone app includes a task that targets attention directed to substance-related cues while the other app includes a similar task that does not target attention in this way. Neither the participants nor the staff members will know which condition the participant has been randomly assigned to. Participants will be informed of the assigned condition by study staff after the completion of the study. In most prior studies, attention training has been delivered on a desktop computer in a laboratory setting. Initial research has shown that attention training can be used in real-world settings using hand-held devices such as smartphones.

ELIGIBILITY:
Inclusion Criteria:

* Able to read and write in English fluently and complete study evaluations
* 6-week availability to participate in the study
* Willing and able to answer questions on smartphones up to 4 times daily for about 10 minutes each time.
* On Suboxone (or methadone if recruitment does not progress as planned) for at least one month (verified by urine drug test- unless using transdermal patch because 1/3 of patients using the patch will not show positive urine screen; and verified by opioid replacement therapy-provider)"
* Meet DSM-5 criteria for opioid use disorder

Exclusion Criteria:

* Use (outside of prescription) for drugs that negatively interact with one another
* Meet severe DSM-5 criteria for current substance use disorders other than opioids, nicotine or cannabis (e.g., current stimulant use disorder) and have used that substance within the past 30 days based on self-report or a positive urine drug test
* Severe psychiatric conditions
* Color blindness and/or uncorrected defective vision

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-08-04 (Actual); Study Completion 2023-06-17 (Actual)

PRIMARY OUTCOMES:
Modified System Usability Scale scores overall and comparisons between study conditions | Post-two-week intervention period
  Seven-point Likert scale items regarding the usability and acceptability of the app (higher score indicates greater usability and acceptability). Higher scores indicate greater usability and acceptability. The attentional bias retraining and control training conditions will also be compared on usability and acceptability scores.
Completion of daily assessments and attendance at study appointments. | Two-week intervention period
  Completion of a high percentage of smartphone assessments and attendance at appointments will show feasibility. Completion of 75% of assessments and attendance at 75% of study appointments will indicate feasibility.
Change in attentional bias (AB) | Two-week intervention period
  Determine if attentional bias retraining reduces attentional bias for opioids compared to a control training condition. Reaction times from both the Visual probe (VP) task and the drug Stroop task will be examined to assess change in AB across time points.

SECONDARY OUTCOMES:
Change in craving levels | Two-week intervention period
  Assess whether attentional bias retraining (ABR) reduces opioid craving to a greater extent than a control training condition based on self-report. Will be examined at each appointment and during the 2-week intervention on the smartphone app. The 14-item Heroin Craving Questionnaire-Short Form (HCQ-SF-14) will be used to measure current heroin/opioid urges at lab appointments, and two questions rated on 6-point Likert scales will be asked after every trial during the smartphone training period about participants current liking and wanting for opioids.
Change in opioid use | Two-week intervention period
  Assess whether attentional bias retraining is associated with less opioid use during the training period than a control training condition based on self-report and urinalysis
Change in pain levels | Two-week intervention period
  The Brief Pain Inventory Short Form (BPI-SF) will be used to measure levels of self-reported pain pre- and post-intervention. Participants will be asked to report daily pain levels during the 2-week intervention period. Self reported pain with the Brief Pain Inventory (BPI)-SF: Self-report questionnaire used to assess the severity of pain and the impact of pain on daily functions. There are 9 items asking participant to rate the worst, least, average, and current pain intensity. Participants are also asked to list current treatments and the perceived effectiveness, and asked to rate the degree that pain interferes with general activity, mood, walking ability, normal work, relations with other persons, sleep, and enjoyment of life on a 10-point scale. The researchers will also ask participants to rate current pain levels, if participants have sought any relief from pain, and what was used to relieve the pain.
Durability of retraining effect on attentional bias | 1-month-follow-up
  Examine the durability of any retraining effects on attentional bias compared to control training at 1-month follow-up. Reaction times from both the visual probe (VP) task and the drug Stroop task will be examined.
Durability of retraining effect on craving | 1-month-follow-up
  Examine the durability of any retraining effects on self-reported craving compared to control training at 1-month follow-up. The 14-item Heroin Craving Questionnaire-Short Form (HCQ-SF-14) will be used to measure current heroin/opioid urges.
Durability of retraining effect on opioid use | 1-month-follow-up
  Examine the durability of any retraining effects on opioid use compared to control training at 1-month follow-up based on self-report and urinalysis.
Durability of retraining effect on pain levels | 1-month-follow-up
  Examine the durability of any retraining effects on self-reported pain compared to control training, measured with The Brief Pain Inventory Short Form (BPI-SF)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Leeman, PhD, Principal Investigator — University of Florida
Locations (1):
- EDGE Laboratory, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No